CLINICAL TRIAL: NCT00449254
Title: A Phase 2a Randomized, Double-Blind, Placebo Controlled, Parallel Group, Safety and Efficacy Study of Oleoyl-Estrone (MP-101) in Male Obese Adults.
Brief Title: Phase 2a Randomized, Double-Blind Study of Oleoyl-Estrone in Male Morbidly Obese Adults
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Manhattan Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAN-OE-US-04
Expanded Access: Available
Record Dates: First submitted 2007-03-16; First posted 2007-03-20 (Estimated); Last update posted 2007-06-05 (Estimated); Status verified 2007-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — oleoyl-estrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: oleoyl-estrone (MP-101)

SUMMARY:
Multi-center, multiple-dose, randomized, double-blind, three-arm, placebo-controlled study of fixed-dose repeated oral dosing for 30 days of 10 mg and 30 mg MP-101 and placebo in obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to provide signed informed consent.
* Subject is a male and is between 18-60 years of age.
* Subject is obese as defined as a BMI of 40 - 55.
* Subject is reasonably healthy and have a reasonably acceptable medical history
* Subject has a stable weight for the past 30 days per subject report.
* Subject who has at least one factor of the metabolic
* Subject exhibits stable behavior patterns with regard to smoking and exercise
* Subject can read, speak and write the English language and agrees to follow study procedures.

Exclusion Criteria:

* Subjects who have received any investigational medication within 3 months prior to administration of study drug
* Subjects with confirmed positive results of UDS or Alcohol
* Subjects who are unwilling to return to the clinical research center on specified days during the treatment periods.
* Subjects who have taken exclusionary medication
* Subjects with any clinically significant laboratory abnormality or illness which, in the opinion of the Investigator, would contraindicate study participation
* Subjects who have a history of testing positive for Hepatitis B virus, Hepatitis C virus, or HIV.
* Subject has been involved in a formal or informal (self-imposed) diet regimen within the last 30 days.
* Subject has a confirmed diagnosis or history of cancer, with the exception of nonmelanoma skin cancer.
* Subject is otherwise unsuitable for the study, in the opinion of the investigator.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2006-10

PRIMARY OUTCOMES:
To evaluate the safety and tolerability

SECONDARY OUTCOMES:
To evaluate the preliminary efficacy

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - St. Luke's-Roosevelt Hospital, New York, New York
  - Research Across America, Dallas, Texas
  - Jean Brown Research, Salt Lake City, Utah